CLINICAL TRIAL: NCT02870049
Title: A RCT of Outreach and Inreach Strategies for Boosting CRC Screening in a Federally-Qualified Health Center
Brief Title: Study to Increase Colorectal Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Samir Gupta, Associate Professor of Clinical Medicine, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 20153270; U54132379 (Other: NCI)
Record Dates: First submitted 2016-08-08; First posted 2016-08-17 (Estimated); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: early detection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Inreach strategy (Experimental): This consists of a community health worker-delivered in clinic education regrading CRC screening with a fecal immunochemical test (FIT) kit, and telephone reminders.
  Interventions: Behavioral: Inreach strategy
- Outreach strategy (Experimental): This consists of mailed invitations to complete screening with an enclosed fecal immunochemical test (FIT) kit and telephone reminders.
  Interventions: Behavioral: Outreach strategy
- Both Inreach and Outreach strategies (Experimental): This is a combination of the above two strategies: Inreach and Outreach combined.
  Interventions: Behavioral: Both Inreach and Outreach strategies
- Usual care (Active Comparator): Usual care in the clinic using the fecal immunochemical test (FIT) kit.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Inreach strategy — Inreach strategy: In clinic education and delivery of fecal immunochemical test (FIT) kit
  Arms: Inreach strategy
Behavioral: Outreach strategy — Outreach strategy: Mailed fecal immunochemical test (FIT) kit and telephone reminders
  Arms: Outreach strategy
Behavioral: Both Inreach and Outreach strategies — Both Inreach and Outreach strategies: Both In clinic education and delivery of fecal immunochemical test (FIT) kit and Mailed fecal immunochemical test (FIT) kit and telephone reminders
  Arms: Both Inreach and Outreach strategies
Behavioral: Usual care — Usual care: FIT kit delivery as part of usual care
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether inreach and outreach strategies will be superior to usual care, and combination of both will be superior to either strategy alone.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) screening saves lives, but screening rates are low among underserved populations, particularly Latinos. The screening rate in the predominantly Latino population served by San Ysidro Health Center (SYHC, a Federally Qualified Health Center (FQHC)), is just 31%, similar to that reported for Latinos nationally, but lower than the overall national average of 65%. Previous research has demonstrated that inreach interventions at point of medical care such as patient navigation after screening referral, and outreach outside of usual medical care (such as with mailed invitations) can increase screening rates among underserved populations. However, since these have undergone limited evaluation among low income predominantly Spanish-speaking Latinos, it is unclear which approach is best, and whether implementing both approaches would be synergistic for optimizing screening rates. We hypothesize that two culturally and linguistically tailored interventions: a) an inreach strategy (IR, consisting of community health worker-delivered in clinic education regarding CRC screening and other components), and b) an outreach strategy (OS, consisting of mailed invitations to complete screening with an enclosed fecal immunochemical test (FIT) and telephone reminders) can substantially increase screening, and further, that the two interventions together will be substantially better than either alone. To test these hypotheses, we propose a randomized trial comparing usual care, IR, OS, and IR+OS for CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 50 to 75 years,
* One or more SYHC visits in the last year,
* Not uptodate with CRC screening

Exclusion Criteria:

* Individuals with personal history of CRC or colorectal polyps

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Gupta, MD, Principal Investigator — University of California, San Diego; Sheila Castaneda, PhD, Principal Investigator — San Diego State University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inreach Strategy | Outreach Strategy | Both Inreach and Outreach Strategies | Usual Care
Started | 168 | 171 | 167 | 167
Completed | 167 | 171 | 166 | 167
Not Completed | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inreach Strategy | Outreach Strategy | Both Inreach and Outreach Strategies | Usual Care | Total
Number analyzed (Participants) | 167 | 171 | 166 | 167 | 671
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (6.5) | 60.0 (7.1) | 60.0 (6.5) | 60.1 (6.3) | 59.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 86 | 86 | 86 | 343
  Male | 82 | 85 | 80 | 81 | 328
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 167 | 171 | 166 | 167 | 671
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 167 | 171 | 166 | 167 | 671

OUTCOME MEASURES:

1. Primary Outcome: Screening Completion Rate
Description: Completion of any colorectal cancer screening test (FIT, sigmoidoscopy or colonoscopy)
Time Frame: 23 months
Measure: Count of Participants; unit: Participants
Arm/Group | Inreach Strategy | Outreach Strategy | Both Inreach and Outreach Strategies | Usual Care
Number analyzed (Participants) | 167 | 171 | 166 | 167
Participants | 46 | 88 | 132 | 131

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Inreach Strategy | Outreach Strategy | Both Inreach and Outreach Strategies | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/171 | 0/167 | 0/167
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/171 | 0/167 | 0/167
Other Adverse Events (participants affected / at risk) | 0/168 | 0/171 | 0/167 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02870049/Prot_SAP_000.pdf